CLINICAL TRIAL: NCT01064310
Title: A Randomised Double-blind Cross-over Patient Preference Study of Pazopanib Versus Sunitinib in Treatment naïve Locally Advanced or Metastatic Renal Cell Carcinoma.
Brief Title: Patient Preference Study of Pazopanib Versus Sunitinib in Advanced or Metastatic Kidney Cancer
Acronym: PISCES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 113046
Record Dates: First submitted 2010-02-04; First posted 2010-02-08 (Estimated); Results first posted 2012-08-23 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Carcinoma, Renal Cell
Keywords: renal cell carcinoma; Votrient; cancer; pazopanib; patient preference; quality of life
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms; Patient Preference | interventions — pazopanib; Sunitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- pazopanib followed by sunitinib (Experimental): 800mg pazopanib orally for 10 weeks followed by 50mg sunitinib orally for 10 weeks
  Interventions: Drug: pazopanib; Drug: sunitinib
- sunitinib followed by pazopanib (Experimental): 50mg sunitinib orally for 10 weeks followed by 800mg pazopanib orally for 10 weeks
  Interventions: Drug: pazopanib; Drug: sunitinib

INTERVENTIONS:
Drug: pazopanib — oral anti-angiogenic treatment
  Other Names: Votrient
Drug: sunitinib — oral anti-angiogenic treatment
  Other Names: Sutent

SUMMARY:
This is a randomised, double-blind, cross-over study of pazopanib versus sunitinib in patients with locally advanced or metastatic renal cell carcinoma (mRCC) who have received no prior systemic therapy for advanced or metastatic RCC. Approximately 160 eligible patients will be stratified based on the ECOG performance status (0 vs. 1) and number of metastatic sites of disease (0 and 1 vs. >=2). The study consists of two treatment periods of 10 weeks with a 2-week wash-out period between the two treatment periods. Patients will receive pazopanib and sunitinib treatment sequentially in a double-blinded fashion. The primary objective of the study is to assess how the tolerability and safety differences between pazopanib and sunitinib translate into patient preference, defined by the patient's stated preference for which drug they may prefer to continue treatment with at end of study. The secondary objectives are to evaluate the reason for patient preference as assessed by a patient preference questionnaire; to evaluate fatigue as assessed by FACIT-Fatigue and quality of life as assessed by EuroQoL EQ-5D; to evaluate dose modifications and time to dose modification; and to evaluate safety.

DETAILED DESCRIPTION:
This is a randomised, double-blind, cross-over study to evaluate the patient preference of pazopanib versus sunitinib in patients with locally advanced or metastatic RCC who have received no prior systemic therapy for advanced or metastatic RCC. Approximately 160 eligible patients will be stratified based on the ECOG performance status (0 vs. 1) and number of metastatic sites of disease (0 and 1 vs. 2+).

The study consists of two 10-weeks treatment periods with a two-week wash-out period between the treatment periods. Patients will receive pazopanib and sunitinib treatment sequentially. At the end of the second treatment period, patient preference and disease assessment are evaluated and the patients are unblinded. Further treatment is at the discretion of the physician. Further treatment with pazopanib is available within the study. Patients requiring other treatments will complete the study at this point.

Patients will be randomized in a 1:1 ratio to receive blinded (overencapsulated) study drug: either 800mg pazopanib orally for 10 weeks followed by 50mg sunitinib orally for 10 weeks or 50mg sunitinib orally for 10 weeks followed by 800mg pazopanib orally for 10 weeks. A two-week washout period will separate the treatment periods (the medical monitor should be consulted if ongoing AEs need to be resolved and the wash-out period needs to be extended). The regimen for sunitinib is 4 weeks of treatment followed by 2 weeks off treatment. To maintain the double-blind during the two weeks off drug for patients on sunitinib ('Treatment Holiday'), patients will be taking matching placebo. No study drug will be taken during the wash-out period in either arm.

Following the two-week wash-out period and disease assessment, all patients are planned to cross over to the second treatment. Patients will be informed of their disease assessment result and any patient that wishes to come off study at this point due to a very significant response, defined as more than a 50% reduction in tumour size (or complete response if non-measurable disease), will have the option to be unblinded to continue with whichever treatment they were on, however each patient case will need to be discussed with the medical monitor prior to unblinding. Patients who were on sunitinib will leave the study and continue treatment outside the study. Patients who were on pazopanib will continue on pazopanib within the pazopanib open-label part of the study. Conversely, should a patient have a very significant response and wish to cross over or complete the study, this must be documented in the patients notes.

Patients crossing over with progressive disease will follow the same visit schedule and assessments and investigators will have the option for these patients to be unblinded or not. The patients' preference will be collected and analysed but will not contribute to the primary, but an exploratory analysis because of the bias caused by progressing on the first treatment. Even if unblinded, patients may continue to receive the second treatment and may receive open label pazopanib after the second treatment within the study if they did not progress on pazopanib.

Patients who withdraw from treatment due to unacceptable toxicity or progression during the first treatment period will cross-over directly to the second treatment following a 2-week wash-out period.

Actual further treatment at the end of the study will be at the discretion of the investigator taking into account both disease assessments results, laboratory results and the patient preference. Choice and rationale for continuing treatment will be documented.

Patients who did not progress on pazopanib and who prefer to continue with pazopanib may continue on pazopanib and will be followed up for safety until the patient comes off pazopanib due to disease progression, toxicity, death or patient choice, which ever is the earliest.

Those patients that may benefit from further treatment with sunitinib for the same reasons as above will receive it off study and will not be followed up, as will patients who receive any other treatment.

Patients are permitted to receive supportive care throughout the study including transfusion of blood and blood products, treatment with antibiotics, anti-emetics, anti-diarrhoeal agents, analgesics, erythropoietin or bisphosphonates, when appropriate. The study treatment will continue until the end of the two treatment periods or unacceptable toxicity or consent withdrawal or death, whichever occurs first.

The patient preference will be ascertained prior to the second disease assessment result being shared with the patient to avoid bias.

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide written informed consent prior to performance of any study-specific procedures or assessments and must be willing to comply with treatment and follow up. Procedures conducted as part of the patient's routine clinical management (e.g. blood count, imaging study) and obtained prior to signing of informed consent may be utilised for screening or baseline purposes provided these procedures are conducted as specified in the protocol.
* Received no prior systemic therapy (including interleukin-2, interferon-alpha, chemotherapy, bevacizumab, mTOR inhibitor, sunitinib, sorafenib or other VEGF TKI) for advanced or metastatic RCC. Patients who received adjuvant treatment with a cancer vaccine are eligible.
* Locally advanced (defined as disease not amenable to curative surgery or radiation therapy) or metastatic renal cell carcinoma of any histology (equivalent to Stage IV RCC according to AJCC staging). Patients with non-measurable disease are allowed if metastatic disease can be confirmed.
* ECOG PS of 0 or 1
* Age >= 18 years
* A female is eligible to enter and participate in this study if she is of:

Non-childbearing potential (i.e. physiologically incapable of becoming pregnant) Childbearing potential, including any female who has had a negative serum pregnancy test within two weeks prior to the first dose of study treatment, preferably as close to the first dose as possible and agrees to use adequate contraception.

* Adequate organ system functions
* Total serum calcium concentration <12.0mg/dL
* Left ventricular ejection fraction (LVEF) >=lower limit of institutional normal (LLN) as assessed by echocardiography (ECHO) or multigated acquisition (MUGA) scan. The same modality used at baseline must be applied for subsequent evaluations.
* Patient is able to swallow and retain oral tablets

Exclusion Criteria:

* Poor MSKCC risk group
* History of another malignancy. Note: Patients who have had another malignancy and have been disease-free for 3 years or patients with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible.
* History or clinical evidence of central nervous system (CNS) metastases.

Note: Patients who have previously-treated CNS metastases (surgery +/- radiotherapy, radiosurgery, or gamma knife) and meet all 3 of the following criteria are eligible:

* Are asymptomatic,
* Have had no evidence of active CNS metastases for >=6 months prior to enrolment ,
* Have no requirement for steroids or enzyme-inducing anticonvulsants (EIAC).
* Any clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding or affect absorption of investigational product including, but not limited to:
* Malabsorption syndrome
* Major resection of the stomach or small bowel that could affect the absorption of study drug
* Active peptic ulcer disease
* Inflammatory bowel disease
* Ulcerative colitis, or other gastrointestinal conditions with increased risk of perforation
* History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment.
* Presence of uncontrolled infection.
* Corrected QT interval (QTc) >480 msecs using Bazett's formula
* History of one or more of the following cardiovascular conditions within the past 6 months:
* Cardiac angioplasty or stenting
* Myocardial infarction
* Unstable angina
* Coronary artery bypass graft surgery
* Symptomatic peripheral vascular disease
* Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
* Poorly controlled hypertension (defined as systolic blood pressure (SBP) of > 150mmHg or diastolic blood pressure (DBP) of > 90mmHg) at baseline.

Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. Blood pressure must be re-assessed on two occasions that are separated by a minimum of 1 hour within a visit. The mean SBP/DBP values from each blood pressure assessment must be <=150/90mmHg in order for a patient to be eligible for the study.

- History of cerebrovascular accident (CVA) including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.

Note: Patients with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible.

* Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major).
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels.
* Evidence of active bleeding or bleeding diathesis.
* Significant haemoptysis within 6 weeks prior to first dose of study drug.
* Any serious and/or unstable pre-existing medical, psychiatric, or other conditions that could interfere with patient's safety, obtaining informed consent or compliance to the study.
* Use any prohibited medications within 14 days of the first dose of study medication.
* Use of an investigational agent, including an investigational anti-cancer agent, within 28 days or 5 half-lives, whichever is longer, prior to the first dose of study drug.
* Radiation therapy, surgery or tumour embolisation within 14 days prior to the first dose of study treatment.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib or sunitinib.
* Pregnant or lactating female Female patients who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2010-05-17 (Actual); Primary Completion 2011-10-19 (Actual); Study Completion 2015-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (50):
- Finland (6):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Joensuu
  - Novartis Investigative Site, Lahti
  - Novartis Investigative Site, Seinäjoki
  - Novartis Investigative Site, Turku
  - Novartis Investigative Site, Vaasa
- France (14):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Colmar
  - Novartis Investigative Site, Hyères
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Priest-en-Jarez
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Villejuif
- Germany (9):
  - Novartis Investigative Site, Ravensburg, Baden-Wurttemberg
  - Novartis Investigative Site, Fürth, Bavaria
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Goslar, Lower Saxony
  - Novartis Investigative Site, Aachen, North Rhine-Westphalia
  - Novartis Investigative Site, Bonn, North Rhine-Westphalia
  - Novartis Investigative Site, Neuss, North Rhine-Westphalia
  - Novartis Investigative Site, Mainz, Rhineland-Palatinate
  - Novartis Investigative Site, Berlin, State of Berlin
- Italy (11):
  - Novartis Investigative Site, Lecce, Apulia
  - Novartis Investigative Site, Meldola (FC), Emilia-Romagna
  - Novartis Investigative Site, Aviano (PN), Friuli Venezia Giulia
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Bergamo, Lombardy
  - Novartis Investigative Site, Monza, Lombardy
  - Novartis Investigative Site, Pavia, Lombardy
  - Novartis Investigative Site, Taormina, Sicily
  - Novartis Investigative Site, Lido Di Camaiore (LU), Tuscany
  - Novartis Investigative Site, Pisa, Tuscany
  - Novartis Investigative Site, Chieti
- United Kingdom (10):
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Bournemouth
  - Novartis Investigative Site, Cottingham
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Norwich
  - Novartis Investigative Site, Plymouth
  - Novartis Investigative Site, Preston
  - Novartis Investigative Site, Shrewsbury
  - Novartis Investigative Site, Wolverhampton

REFERENCES:
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] Oudard S, Benhamouda N, Escudier B, Ravel P, Tran T, Levionnois E, Negrier S, Barthelemy P, Berdah JF, Gross-Goupil M, Sternberg CN, Bono P, Porta C, De Giorgi U, Parikh O, Hawkins R, Highley M, Wilke J, Decker T, Tanchot C, Gey A, Terme M, Tartour E. Decrease of Pro-Angiogenic Monocytes Predicts Clinical Response to Anti-Angiogenic Treatment in Patients with Metastatic Renal Cell Carcinoma. Cells. 2021 Dec 22;11(1):17. doi: 10.3390/cells11010017. PMID 35011579
- [Derived] Lai JS, Beaumont JL, Diaz J, Khan S, Cella D. Validation of a short questionnaire to measure symptoms and functional limitations associated with hand-foot syndrome and mucositis in patients with metastatic renal cell carcinoma. Cancer. 2016 Jan 15;122(2):287-95. doi: 10.1002/cncr.29655. Epub 2015 Oct 12. PMID 26457466
- [Derived] Escudier B, Porta C, Bono P, Powles T, Eisen T, Sternberg CN, Gschwend JE, De Giorgi U, Parikh O, Hawkins R, Sevin E, Negrier S, Khan S, Diaz J, Redhu S, Mehmud F, Cella D. Randomized, controlled, double-blind, cross-over trial assessing treatment preference for pazopanib versus sunitinib in patients with metastatic renal cell carcinoma: PISCES Study. J Clin Oncol. 2014 May 10;32(14):1412-8. doi: 10.1200/JCO.2013.50.8267. Epub 2014 Mar 31. PMID 24687826

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were169 participants randomized and one participant randomized in error with no data available
Groups:
- Sunitinib 50 mg Followed by Pazopanib 800 mg: Period 1: Participants received 4 overencapsulated capsules of sunitinib, each containing 12.5 milligrams (mg) of sunitinib, once daily (OD) orally for 4 weeks, followed by 2 weeks off treatment (matching placebo capsules to maintain blind), followed by 50 mg (4 x 12.5 mg) OD orally for 4 weeks. Period 1 was followed by a 2-week wash-out period in which no treatment was given. Period 2: Participants received 4 overencapsulated tablets of pazopanib, each containing 200 mg of pazopanib, OD orally for 10 weeks. Study drugs were taken without food at least one hour before or two hours after a meal. The capsules were swallowed whole and not crushed or broken. The time of day the study drugs were taken remained relatively constant.
- Pazopanib 800 mg Followed by Sunitinib 50 mg: Period 1: Participants received 4 overencapsulated tablets of pazopanib, each containing 200 mg of pazopanib, OD orally for 10 weeks. Period 1 was followed by a 2-week wash-out period in which no treatment was given. Period2: Participants received 4 overencapsulated capsules of sunitinib, each containing 12.5 mg of sunitinib, OD orally for 4 weeks, followed by 2 weeks off treatment (matching placebo capsules to maintain blind), followed by 50 mg (4 x 12.5 mg) OD orally for 4 weeks. Study drugs were taken without food at least one hour before or two hours after a meal. The capsules were swallowed whole and not crushed or broken. The time of day the study drugs were taken remained relatively constant.
- Open Label Pazopinib: To provide continued access to treatment
Period: Period 1
Arm/Group | Sunitinib 50 mg Followed by Pazopanib 800 mg | Pazopanib 800 mg Followed by Sunitinib 50 mg | Open Label Pazopinib
Started | 82 | 86 | 0
Completed | 68 | 68 | 0
Not Completed | 14 | 18 | 0
Not completed — Adverse Event | 7 | 10 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0
Not completed — Lack of Efficacy | 3 | 5 | 0
Not completed — Entered Open-label Period | 1 | 1 | 0
Period: Period 2
Arm/Group | Sunitinib 50 mg Followed by Pazopanib 800 mg | Pazopanib 800 mg Followed by Sunitinib 50 mg | Open Label Pazopinib
Started | 68 | 68 | 0
Completed | 64 | 62 | 0
Not Completed | 4 | 6 | 0
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Entered Open-label Period | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 4 | 0
Period: Open Label Pazopinib
Arm/Group | Sunitinib 50 mg Followed by Pazopanib 800 mg | Pazopanib 800 mg Followed by Sunitinib 50 mg | Open Label Pazopinib
Started | 0 | 0 | 84
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 84
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 12
Not completed — Lack of Efficacy | 0 | 0 | 51
Not completed — Physician Decision | 0 | 0 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sunitinib 50 mg Followed by Pazopanib 800 mg | Pazopanib 800 mg Followed by Sunitinib 50 mg | Total
Number analyzed (Participants) | 82 | 86 | 168
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.1 (9.56) | 62.2 (11.35) | 62.2 (10.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 25 | 55
  Male | 52 | 61 | 113
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 1 | 0 | 1
  Asian-Central/South Asian Heritage | 1 | 0 | 1
  White | 74 | 83 | 157
  Missing | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Preference for Pazopanib Versus Sunitinib as Assessed by the Patient Preference Questionnaire (PPQ)
Description: The PPQ is used to measure participants' preference for pazopanib or sunitinib for renal cell carcinoma management and is used to determine a participant's preference for 1 of the 2 drugs given in the 2 double-blind treatment periods. Participants were asked to select 1 of the following: 1. prefer the drug taken as the first treatment; 2. prefer the drug taken as the second treatment; or 3, no preference. Those participants who indicated a preference were asked to select the factors that had an influence on their treatment preference, as well as the most important reason for their preference.
Time Frame: End of treatment of both study drugs (maximum of 22 weeks)
Population: Modified-Intent-to-Treat (mITT) Population (used for the primary analysis): participants who received at least one dose of study treatment from each treatment period and who did not have documented progressive disease (PD) at the end of Treatment Period 1 and completed the patient preference questionnaire.
Measure: Number; unit: participants
Arm/Group | Sunitinib 50 mg Followed by Pazopanib 800 mg | Pazopanib 800 mg Followed by Sunitinib 50 mg
Number analyzed (Participants) | 60 | 54
participants
  Sunitinib | 19 | 6
  Pazopanib | 37 | 43
  No preference | 4 | 5
Statistical Analysis 1: Comparison: Sunitinib 50 mg Followed by Pazopanib 800 mg vs Pazopanib 800 mg Followed by Sunitinib 50 mg; Test type: Superiority or Other; p < 0.001, Prescotts test — The p value indicates the difference in preference for pazopanib versus sunitinib treatment; Percentage of participants = 49.26, 90% CI 2-sided [37.0 to 61.5] — The estimated value indicates the difference in the percentage of participants who preferred pazopanib versus sunitinib. This difference is adjusted for sequence

2. Primary Outcome: Number of Participants Answering "Yes," "no," or Not Applicable (N/A) to the Question of Whether the Indicated Factors Influenced Their Preference for Sunitinib or Pazopanib Treatment as Assessed by the Patient Preference Questionnaire
Description: as for outcome 1
Time Frame: End of treatment of both study drugs (maximum of 22 weeks)
Population: mITT Population. Responses to some categories of the PPQ may be missing for some participants.
Measure: Number; unit: participants
Groups:
- Sunitinib: Participants received 4 overencapsulated capsules of sunitinib (either in Period 1 or Period 2), each containing 12.5 mg of sunitinib, OD orally for 4 weeks, followed by 2 weeks off treatment (matching placebo capsules to maintain blind), followed by 50 mg (4 x 12.5 mg) OD orally for 4 weeks. Study drug was taken orally OD without food at least one hour before or two hours after a meal. The capsules were swallowed whole and not crushed or broken. The time of day the study drug was taken remained relatively constant.
- Pazopanib: Participants received 4 overencapsulated tablets of pazopanib (either in Period 1 or Period 2), each containing 200 mg of pazopanib, OD orally for 10 weeks. Study drug was taken orally OD without food at least one hour before or two hours after a meal. The capsules were swallowed whole and not crushed or broken. The time of day the study drug was taken remained relatively constant.
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 25 | 80
participants
  Fatigue had less impact on life, Yes | 12 | 47
  Fatigue had less impact on life, No | 8 | 26
  Fatigue had less impact on life, not applicable (N | 5 | 6
  Soreness in hands/feet had less impact, Yes | 6 | 30
  Soreness in hands/feet had less impact, No | 7 | 22
  Soreness in hands/feet had less impact, NA | 12 | 28
  Soreness in mouth/throat had less impact, Yes | 6 | 32
  Soreness in mouth/throat had less impact, No | 8 | 25
  Soreness in mouth/throat had less impact, NA | 11 | 23
  Loss of appetite had less impact, Yes | 10 | 28
  Loss of appetite had less impact, No | 8 | 28
  Loss of appetite had less impact, NA | 7 | 22
  Change in hair color had less impact, Yes | 5 | 9
  Change in hair color had less impact, No | 11 | 51
  Change in hair color had less impact, NA | 9 | 20
  Nausea/vomiting had less impact, Yes | 11 | 32
  Nausea/vomiting had less impact, No | 7 | 30
  Nausea/vomiting had less impact, NA | 7 | 17
  Diarrhea had less impact, Yes | 16 | 21
  Diarrhea had less impact, No | 5 | 44
  Diarrhea had less impact, NA | 4 | 15
  Pain in stomach area had less impact, Yes | 9 | 23
  Pain in stomach area had less impact, No | 4 | 30
  Pain in stomach area had less impact, NA | 12 | 27
  Changes in food tastes had less impact, Yes | 5 | 44
  Changes in food tastes had less impact, No | 14 | 23
  Changes in food tastes had less impact, NA | 6 | 12
  Quality of life better, Yes | 15 | 65
  Quality of life better, No | 6 | 12
  Quality of life better, NA | 4 | 2
  Other, Yes | 5 | 14
  Other, No | 0 | 0
  Other, NA | 20 | 66

3. Secondary Outcome: Change From Period Baseline (BL) in Fatigue as Assessed by the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score
Description: Change from period (P) BL is computed as participants' (par.) average post-BL fatigue score within each P minus their P-specific BL score. P 1 BL is the P 1 Pre-Dose assessment; P 2 BL is the wash-out assessment. Crossover analyses compared par. average scores on each treatment, adjusting for sequence. FACIT-Fatigue Scale: overall score (0 to 52)=the sum of scores for 13 questions. For each question, par. rated their condition for the past week on a 5-point scale: 0 (not at all) to 4 (very much). A high score indicates low fatigue. A negative change from BL represents a worsening of condition.
Time Frame: Day 1 (Period [P] 1 Pre-dose); Weeks 2, 4, 6, 8, and 10 of P 1; during 2-week Wash-out Period (Study Weeks 11 and 12); Weeks 2, 4, 6, and 8 of P 2 (Study Weeks 14, 16, 18, 20, and 22, respectively); End of Study (Week 10 of P 2 [Study Week 22])
Population: Safety-Randomized Study Population: participants who received at least one dose of either drug regardless of treatment period. Participants who received mixed treatment within a period were excluded. Only those participants contributing data at the indicated time points were evaluated.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sunitinib 50 mg Followed by Pazopanib 800 mg | Pazopanib 800 mg Followed by Sunitinib 50 mg
Number analyzed (Participants) | 77 | 79
Scores on a scale
  Period 1 Average; n=77, 79 | -4.4 (7.73) | -4.6 (9.22)
  Period 2 Average; n=63, 65 | -3.6 (7.11) | -7.3 (11.16)

4. Secondary Outcome: Quality of Life as Assessed by the EuroQoL-5 Dimensions (EQ-5D) Thermometer and Utility Scores
Description: The EQ-5D is a participant-answered questionnaire measuring 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ-5D has two separate components: utility score and thermometer score. The EQ-5D total utility score ranges from 0 (worst health state) to 1 (perfect health state); 1 reflects the best outcome. The thermometer score ranges from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Day 1 (Period 1 Pre-dose); during 2-week Wash-out Period (Study Weeks 11 and 12); and End of Study (Week 10 of Period 2 [Study Week 22])
Population: Safety-Randomized Study Population. Participants (par.) who received mixed treatment within a period were excluded. Only those par. contributing data at the indicated time points were evaluated. In some instances, par. may have contributed data for one score, but not the other; thus, the number of par. analyzed reflects the entire population.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sunitinib 50 mg Followed by Pazopanib 800 mg | Pazopanib 800 mg Followed by Sunitinib 50 mg
Number analyzed (Participants) | 80 | 86
Scores on a scale
  Thermometer Score, Day 1; n=74, 79 | 75.7 (17.65) | 74.8 (18.54)
  Thermometer Score, Washout; n=60, 63 | 74.4 (16.76) | 69.8 (19.94)
  Thermometer Score, End of Study; n=51, 45 | 71.3 (16.19) | 65.1 (22.55)
  Utility Score, Day 1; n=76, 81 | 0.7625 (0.25331) | 0.7664 (0.22946)
  Utility Score, Washout; n=61, 67 | 0.8103 (0.20776) | 0.7595 (0.26826)
  Utility Score, End of Study; n=52, 47 | 0.7487 (0.21324) | 0.6325 (0.29635)

5. Secondary Outcome: Time to Dose Modification
Description: For the subset of participants who had a dose modification, time to dose modification was defined as the time from the first dose in each period until the first reduction in dose within a period.
Time Frame: End of second treatment period (maximum of 22 weeks)
Population: Safety-Randomized Study Population. Only those participants who had a dose modification were evaluated.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 30 | 20
weeks | 3.7 [2.7 to 5.9] | 4.0 [2.1 to 6.0]

6. Secondary Outcome: Number of Participants With the Indicated Number of Dose Reductions
Description: Participants are recorded under the treatment they were receiving at the time the dose reduction was reported.
Time Frame: End of second treatment period (maximum of 22 weeks)
Population: Safety-Randomized Study Population. Only those participants who had an dose reduction were evaluated.
Measure: Number; unit: participants
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 30 | 20
participants
  1 | 16 | 8
  2 | 10 | 11
  3 or more | 4 | 1

7. Secondary Outcome: Number of Participants With the Indicated Reason for Receiving a Dose Reduction
Description: Dose reduction of study drug was a stepwise reduction of the dose of the study drug: one less capsule was received at each step reduction. Participants were monitored for approximately 10 to 14 days at each dose level. Participants are recorded under the treatment they were receiving at the time the dose reduction was reported.
Time Frame: End of second treatment period (maximum of 22 weeks)
Population: Safety-Randomized Study Population. Only those participants who had an dose reduction were evaluated. Participants may be counted multiple times for the same "reason" for a dose reduction if the participant had multiple reductions for the same reason.
Measure: Number; unit: participants
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 30 | 20
participants
  Adverse Event | 46 | 33
  Other | 3 | 0

8. Secondary Outcome: Number of Participants With Grade 1 to Grade 5 Adverse Events (AEs)
Description: AEs were graded using the Common Toxicity Criteria from the Cancer Therapy Evaluation Program, Division of Cancer Therapy, National Cancer Institute. Grades: 0 = No AE or within normal limits; 1 = Mild AE; 2 = Moderate AE; 3 = Severe and undesirable AE; 4 = Life-threatening or disabling AE; 5 = Death related to AE.
Time Frame: Baseline to end of study (maximum of 22 weeks)
Population: Safety-Randomized Study Population
Measure: Number; unit: participants
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 148 | 153
participants
  Grade 0 | 0 | 0
  Grade 1 | 20 | 25
  Grade 2 | 57 | 63
  Grade 3 | 58 | 51
  Grade 4 | 11 | 8
  Grade 5 | 1 | 0

9. Secondary Outcome: Number of Participants With the Indicated AEs Leading to Permanent Discontinuation of Study Treatment
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE that spans more than one period is considered to be an AE for each period during which the AE increased in grade. There is only one action with respect to study drug recorded for the whole event. As such, it is not always possible to determine in which study period treatment was discontinued due to the AE.
Time Frame: Baseline to end of study (maximum of 22 weeks)
Population: Safety-Randomized Study Population. Only those participants with adverse events leading to permanent discontinuation of study treatment were evaluated.
Measure: Number; unit: participants
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 38 | 25
participants
  Fatigue | 5 | 3
  Alanine aminotransferase increased | 2 | 4
  Vomiting | 1 | 3
  Aspartate aminotransferase increased | 0 | 3
  Diarrhoea | 1 | 2
  Thrombocytopenia | 3 | 0
  Acute myocardial infarction | 1 | 1
  Asthenia | 2 | 0
  Back pain | 1 | 1
  Dyspnoea | 2 | 0
  Epistaxis | 2 | 0
  Hypertension | 2 | 0
  Nasal congestion | 1 | 1
  Pleural effusion | 2 | 0
  Transient ischaemic attack | 0 | 2
  Atrial flutter | 0 | 1
  Blood potassium decreased | 1 | 0
  Cardiac disorder | 0 | 1
  Cardiac failure | 0 | 1
  Cough | 1 | 0
  Decreased appetite | 1 | 0
  Dizziness | 0 | 1
  Dysgeusia | 0 | 1
  Haematemesis | 0 | 1
  Haematoma | 1 | 0
  Haematuria | 1 | 0
  Haemorrhage intracranial | 1 | 0
  Headache | 1 | 0
  Hepatic function abnormal | 0 | 1
  Hepatotoxicity | 0 | 1
  Infection | 1 | 0
  Infectious peritonitis | 0 | 1
  Influenza | 1 | 0
  Influenza like illness | 1 | 0
  Mucosal inflammation | 1 | 0
  Myocardial ischaemia | 0 | 1
  Nausea | 0 | 1
  Neutropenic infection | 1 | 0
  Ovarian cyst | 1 | 0
  Pain in extremity | 1 | 0
  Palmar-plantar erythrodysaesthesia syndrome | 1 | 0
  Pancytopenia | 1 | 0
  Proteinuria | 0 | 1
  Pyrexia | 1 | 0
  Rash | 0 | 1
  Renal failure | 1 | 0
  Respiratory failure | 0 | 1
  Sinusitis | 1 | 0
  Skin ulcer | 0 | 1
  Spinal cord compression | 0 | 1
  Stomatitis | 1 | 0
  Tooth infection | 1 | 0
  Transaminases increased | 1 | 0
  Urine protein/creatinine ratio decreased | 1 | 0
  Weight decreased | 1 | 0

10. Secondary Outcome: Change From Baseline (BL) in Systolic Blood Pressure (SBP) and Diastolic BP (DBP)
Description: When the heart beats, it contracts and pushes blood through the arteries to the rest of body. This force creates pressure on the arteries called SBP. DBP is the pressure in the arteries when the heart rests between beats. Normal levels: SBP (120 mmHg or less); DBP (80 mmHg or less). Mean change from BL for each assessment week was calculated as the average change from period BL at the specified visits (combining data across P 1 and 2 for Weeks 2 and 6). Study weeks are approximate; participants could have crossed over from P 1 to P 2 at earlier time points than specified in the protocol.
Time Frame: Baseline of Period (P) 1 (Screening); Period 1 Weeks 2 and 6 (Study Weeks 2 and 6); Baseline of Period 2 (Washout=Study Week 12); Period 2 Weeks 2, 6, and 10 (Study Weeks 14, 18, and 22)
Population: Safety-Randomized Study Population. All participants who received sunitinib or pazopanib either during Period 1 or Period 2 were counted in both treatment groups (sunitinib and pazopanib). Only those participants contributing data at the indicated time points were evaluated.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 139 | 147
Millimeters of mercury (mmHg)
  SBP, Week 2; n=139, 147 | 6.3 (15.26) | 7.5 (16.36)
  SBP, Week 6; n=109, 134 | -0.4 (18.65) | 7.5 (17.21)
  SBP, Week 10; n=61, 64 | 4.5 (18.43) | 4.7 (20.45)
  DBP, Week 2; n=139, 147 | 6.5 (9.91) | 6.5 (10.49)
  DBP, Week 6; n=109, 134 | -0.4 (9.48) | 6.9 (10.87)
  DBP, Week 10; n=61, 64 | 3.1 (10.69) | 5.6 (11.44)

11. Secondary Outcome: Change From Baseline (BL) in Heart Rate
Description: Heart rate (HR) is the number of heartbeats per unit of time, typically expressed as beats per minute. HR can vary as the body's need to absorb oxygen and excrete carbon dioxide changes, such as during exercise or sleep. A normal resting HR ranges from 60 to 100 beats per minute. Mean change from BL for each assessment week was calculated as the average change from period BL at the specified visits (combining data across P 1 and 2 for Weeks 2 and 6). Study weeks are approximate; participants could have crossed over from P 1 to P 2 at earlier time points than specified in the protocol.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 137 | 145
Beats per minute
  Week 2, n=137, 145 | -3.1 (12.39) | -2.7 (13.09)
  Week 6, n=106, 131 | 0.8 (11.43) | -3.3 (12.41)
  Week 10, n=60, 64 | -3.8 (13.54) | -1.8 (13.84)

ADVERSE EVENTS:
Groups:
- Sunitinib: Sunitinib
- Pazopanib: Pazopanib
- Open Label Pazopanib: Open Label Pazopanib
Arm/Group | Sunitinib | Pazopanib | Open Label Pazopanib
Serious Adverse Events (participants affected / at risk) | 35/148 | 30/153 | 15/84
Other Adverse Events (participants affected / at risk) | 143/148 | 142/153 | 73/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=148) | Pazopanib (N=153) | Open Label Pazopanib (N=84)
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 3 | 2 | 1
General physical health deterioration (General disorders) | 3 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Performance status decreased (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 1
Biliary sepsis (Infections and infestations) | 0 | 0 | 1
Colonic abscess (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 2 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Neutropenic infection (Infections and infestations) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Lipase abnormal (Investigations) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 2 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 2 | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=148) | Pazopanib (N=153) | Open Label Pazopanib (N=84)
Anaemia (Blood and lymphatic system disorders) | 5 | 4 | 5
Neutropenia (Blood and lymphatic system disorders) | 8 | 6 | 4
Hypothyroidism (Endocrine disorders) | 6 | 6 | 5
Abdominal pain (Gastrointestinal disorders) | 16 | 20 | 11
Abdominal pain upper (Gastrointestinal disorders) | 19 | 7 | 8
Constipation (Gastrointestinal disorders) | 23 | 13 | 10
Diarrhoea (Gastrointestinal disorders) | 49 | 63 | 45
Dyspepsia (Gastrointestinal disorders) | 23 | 17 | 6
Flatulence (Gastrointestinal disorders) | 5 | 10 | 5
Haemorrhoids (Gastrointestinal disorders) | 10 | 3 | 1
Nausea (Gastrointestinal disorders) | 46 | 50 | 26
Stomatitis (Gastrointestinal disorders) | 22 | 7 | 5
Vomiting (Gastrointestinal disorders) | 26 | 21 | 18
Asthenia (General disorders) | 35 | 26 | 16
Fatigue (General disorders) | 42 | 43 | 25
Mucosal inflammation (General disorders) | 32 | 25 | 6
Pyrexia (General disorders) | 10 | 5 | 1
Jaundice (Hepatobiliary disorders) | 8 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 5
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 6
Urinary tract infection (Infections and infestations) | 4 | 5 | 5
Alanine aminotransferase increased (Investigations) | 5 | 9 | 7
Blood creatinine increased (Investigations) | 5 | 2 | 5
Blood thyroid stimulating hormone increased (Investigations) | 2 | 0 | 5
Weight decreased (Investigations) | 7 | 9 | 9
Decreased appetite (Metabolism and nutrition disorders) | 30 | 32 | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 11 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 13 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 9 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 5 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 9 | 2
Dysgeusia (Nervous system disorders) | 40 | 25 | 12
Headache (Nervous system disorders) | 17 | 22 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 6 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 12 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15 | 8 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 11 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 14 | 6 | 6
Erythema (Skin and subcutaneous tissue disorders) | 5 | 8 | 3
Hair colour changes (Skin and subcutaneous tissue disorders) | 19 | 26 | 9
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 39 | 27 | 11
Rash (Skin and subcutaneous tissue disorders) | 17 | 13 | 10
Skin depigmentation (Skin and subcutaneous tissue disorders) | 6 | 8 | 1
Hypertension (Vascular disorders) | 37 | 32 | 13

LIMITATIONS AND CAVEATS:
The study remained open to allow subjects currently on treatment continued access to treatment with open label pazopanib.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.